CLINICAL TRIAL: NCT04125433
Title: Use of Information Technology to Support Integration of Social Determinant of Health Services to Reduce Avoidable Emergency Department Visits
Brief Title: IT to Support Integration of Social Determinant of Health Services to Reduce Avoidable Emergency Department Visits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern New York Rural Behavioral Health Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCBHNPIC
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Mental Health Issue; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: In this study a Medicaid Managed Care Plan will identify up to 400 plan members who have visited an emergency department greater than 6 time in a 12-month period. These individuals will receive enhanced integrated peer care services and will be tracked across health and social service venues using a single IT platform. This study will examine the impact of this intervention on total cost of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medicaid Emergency Department High Utilizers (Experimental): This Arm will include the following individuals
  * Up to 400 Adults age 18 to 65
  * New York State Medicaid Managed Care Members
  * Have utilized emergency department services 6 or more times in a 12-month period
  * Have been assigned to the Pilot Project by their Medicaid Managed Care Plan
  Interventions: Behavioral: Peer Integrated Care Services

INTERVENTIONS:
Behavioral: Peer Integrated Care Services — The project employs a two level intervention to include Peer Support Specialist (PSS) and Community Health Advocate (CHA). Contact and engagement with participating members will be through both direct intervention in the emergency department as well as in the community for prevention visits and follow up. Peers and Community Health Advocates will address Behavioral and Social Determinants of Health (SDoH) concerns through a coordinated intervention supported by a common IT Medicaid member tracking platform. This research project will determine the feasibility of deploying a single shared IT platform that will include referral, appointment completion, and intervention outcome data. Project staff will develop a relationship with the members improving member access and engagement with community-based services. The project will determine the impact on total cost of care through redirecting study participants to community resources rather than return visits to the emergency department.

SUMMARY:
Working through regional Accountable Care Organizations (ACO) the sponsor will establish a 2-year pilot project to demonstrate that early recognition and intervention in the various Social Determinant of Health (SDoH) domains can reduce avoidable Emergency Department (ED) visits by high utilizers. The regional ACO's will contract with Medicaid Managed Care Plans to assign traditional high ED utilizing members to the pilot project. Members will be offered enhanced peer facilitated care management services connecting members with available SDoH community based services. Members fitting our eligibility criteria will self-select by way of completing a pilot project consent form.

DETAILED DESCRIPTION:
The project employs a two level intervention to include Peer Support Specialist (PSS) and Community Health Advocate (CHA). Contact and engagement with participating members will be through both direct intervention in the emergency department by Peer Support Specialist (the peer) as well as in the community for prevention visits and follow up by both the peer and Community Health Advocate. These well-positioned Peers and Community Health Advocates will address Behavioral and Social Determinants of Health (SDoH) concerns through a highly coordinated intervention supported by a common IT Medicaid member tracking platform. This research project will determine the feasibility of deploying a single shared IT platform that will include referral, appointment completion, and intervention outcome data. Project staff will develop a trusting relationship with the members and will improve member access and engagement with community-based services. The project will also seek to determine the impact on total cost of care through redirecting study participants to community resources that are more appropriate, and less expensive than return visits to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 65
* New York State Medicaid Managed Care Members
* Have utilized emergency department services 6 or more times in a 12-month period
* Have been assigned to the Pilot Project by their Medicaid Managed Care Plan

Exclusion Criteria:

* Individuals not assigned by a Managed Care Organization meeting the above criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adoption and Use of IT Platform | Months 6, 12, 18, 24
  Change in Number of Participating Agencies That Contribute Data to the IT System
Change in Engagement of Medicaid Member Participants with Peer Integration Care Services | Months 0, 3, 6, 9, 12, 15, 18, 21, 24
  The change in acceptance by Medicaid Members of Peer Integrated Care Services
Change in Total Cost of Care for Participating Members | Month 0, Month 24
  Change in cost trend for participating members. Pre-study vs. study period.

SECONDARY OUTCOMES:
Change in Emergency Room Visits by Participating Members | Month 0, 6, 12,18,24
  Change in rate of Emergency Department utilization by participating members.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cawley, BBA, Principal Investigator — Northern NY Rural Behavioral Health Institute
Locations (1):
- Northern New York Rural Behavioral Health Institute, Saranac Lake, New York, United States

IPD SHARING:
Plan to Share IPD: No